CLINICAL TRIAL: NCT06948448
Title: A Randomized, Open Label, Multicenter, Phase 2 Study to Evaluate the Safety and Efficacy of Two Dose Levels of ONO-4578 With Opdivo® in Combination With mFOLFOX6 and Bevacizumab Versus Standard of Care for First-line Treatment of Non-MSI-H/dMMR, PD-L1 Positive Advanced Colorectal Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Two Dose Levels of ONO-4578 With Opdivo®, in Combination With mFOLFOX6 and Bevacizumab Versus Standard of Care in Participants With Non-MSI-H/dMMR, PD-L1 Positive Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4578-10
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Oxaliplatin; Fluorouracil; Bevacizumab; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A ONO-4578 dose 1 + Opdivo® + SOC (mFOLFOX6 + bevacizumab) (Experimental)
  Interventions: Drug: ONO-4578; Drug: Opdivo®; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin
- Arm B ONO-4578 dose 2 + Opdivo® + SOC (mFOLFOX6 + bevacizumab) (Experimental)
  Interventions: Drug: ONO-4578; Drug: Opdivo®; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin
- Arm C SOC (mFOLFOX6+bevacizumab) (Active Comparator)
  Interventions: Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin

INTERVENTIONS:
Drug: ONO-4578 — ONO-4578 tablets once a day
  Arms: Arm A ONO-4578 dose 1 + Opdivo® + SOC (mFOLFOX6 + bevacizumab); Arm B ONO-4578 dose 2 + Opdivo® + SOC (mFOLFOX6 + bevacizumab)
Drug: Opdivo® — Specified dose on specified days
  Other Names: Nivolumab
  Arms: Arm A ONO-4578 dose 1 + Opdivo® + SOC (mFOLFOX6 + bevacizumab); Arm B ONO-4578 dose 2 + Opdivo® + SOC (mFOLFOX6 + bevacizumab)
Drug: Oxaliplatin — Specified dose on specified days
Drug: 5-Fluorouracil — Specified dose on specified days
Drug: Bevacizumab — Specified dose on specified days
Drug: Leucovorin — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two dose levels of ONO-4578 with Opdivo® when added to mFOLFOX6 and bevacizumab versus SOC as first-line treatment for advanced CRC.

DETAILED DESCRIPTION:
Potential participants will be consented and screened for study eligibility. Eligible participants will be randomized in a 1:1:1 ratio to one of the three study intervention arms. Study intervention will be administered in 28-day treatment cycles and continued until disease progression, intolerable toxicity, Investigator decision or withdrawal of consent by the participant, or termination of the study by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced (locally advanced or metastatic) colorectal cancer not amenable to curative resection
* ECOG Performance Status of 0-1
* No prior systemic treatment for advanced local or mCRC
* Participants whose tumor is positive for PD-L1 expression as determined at a central laboratory

Exclusion Criteria:

* Participants with high microsatellite instability (MSI-High), or mismatch repair deficient (dMMR) tumor
* Participants with BRAF V600E mutation
* Unable to swallow tablets.
* Participants with complication or history of interstitial lung disease, pneumonitis or pulmonary fibrosis
* Participants with an active, known or suspected autoimmune disease.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-02-15 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) per Blinded Independent Central Review (BICR) | From randomization to the end of treatment (Up to 39 months)
  ORR (assessed by BICR per RECIST v1.1) is defined as the proportion of participants with a BOR of confirmed CR or PR. The ORR will be estimated as the number of participants achieving BOR of CR or PR assessed by BICR per RECIST v1.1 divided by the total number of participants.
Number of participants with Adverse Events (AEs) | From first dose to 28 days post last dose
  An AE is any untoward medical occurrence in a patient or clinical study patient, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of participants with Serious Adverse Events (SAEs) | From first dose to 28 days post last dose
  SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in significant disability/incapacity.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  ORR (assessed by site Investigator per RECIST v1.1) is defined as the proportion of participants with a BOR of confirmed CR or PR. The ORR will be estimated as the number of participants achieving BOR of CR or PR assessed by site Investigator per RECIST v1.1 divided by the total number of participants.
Overall Survival (OS) | From randomization to the end of treatment (Up to 39 months)
  OS is defined as the time between the date of randomization and the date of death due to any cause.
Progression-Free Survival (PFS) by BICR | From randomization to the end of treatment (Up to 39 months)
  PFS by BICR is defined as the time from date of randomization to the date of the first documented progressive disease (PD) as determined by BICR per RECIST version 1.1, or the date of death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  PFS by Investigator assessment is defined as the time from date of randomization to the date of the first documented progressive disease (PD) as determined by site Investigator per RECIST version 1.1, or the date of death due to any cause, whichever occurs first.
Best overall response (BOR) by BICR | From randomization to the end of treatment (Up to 39 months)
  BOR is defined as the best response designation, recorded between the start of the study intervention and the date of the initial objectively documented PD per RECIST v1.1 or the date of subsequent anti-cancer therapy, whichever occurs first.
Best overall response (BOR) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  BOR is defined as the best response designation, recorded between the start of the study intervention and the date of the initial objectively documented PD per RECIST v1.1 or the date of subsequent anti-cancer therapy, whichever occurs first.
Duration of response (DOR) by BICR | From randomization to the end of treatment (Up to 39 months)
  DOR is defined as the time between the date of first confirmed CR or PR to the date of the first documented PD per RECIST v1.1 or death due to any cause, whichever occurs first.
Duration of response (DOR) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  DOR is defined as the time between the date of first confirmed CR or PR to the date of the first documented PD per RECIST v1.1 or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) by BICR | From randomization to the end of treatment (Up to 39 months)
  DCR is defined as the percentage of participants whose BOR is determined to be CR, PR, or stable disease (SD).
Disease Control Rate (DCR) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  DCR is defined as the percentage of participants whose BOR is determined to be CR, PR, or stable disease (SD).
Time to Response (TTR) by BICR | From randomization to the end of treatment (Up to 39 months)
  TTR is defined as the time from the date of randomization to the date of first confirmed CR or PR.
Time to Response (TTR) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  TTR is defined as the time from the date of randomization to the date of first confirmed CR or PR.
Maximum percent change in the sum of the diameters of the target lesions by BICR | From randomization to the end of treatment (Up to 39 months)
  In participants who have target lesions at baseline and at least 1 post-baseline imaging evaluation, the maximum percent change in the sum of diameters of target lesions is the percent change at the point of the minimum sum of diameters of the target lesions.
Maximum percent change in the sum of the diameters of the target lesions by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  In participants who have target lesions at baseline and at least 1 post-baseline imaging evaluation, the maximum percent change in the sum of diameters of target lesions is the percent change at the point of the minimum sum of diameters of the target lesions.
Progression-Free Survival of second line therapy (PFS2) by Investigator assessment | From randomization to the end of treatment (Up to 39 months)
  PFS2 is defined as the time from date of randomization to the date of an overall response of PD after subsequent anti-cancer therapy, initiating date of a second subsequent anti-cancer therapy, or date of death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (17):
- United States (7):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Baylor Scott & White Medical Center, Temple, Texas
  - Blue Ridge Cancer Care, Salem, Virginia
- Princess Margaret Cancer Centre- University Health Network, Toronto, Ontario, Canada
- France (4):
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hôpital de la Timone, Marseille, Marseille
  - Hôpital Européen Georges Pompidou, Paris, Paris
  - Hôpital Saint-Antoine, Paris, Paris
- Japan (4):
  - Kobe City Medical Center General Hospital, Hyōgo, Kobe-shi
  - National Hospital Organization Osaka National Hospital, Osaka, Osaka-shi
  - Osaka General Medical Center, Osaka, Osaka-shi
  - Osaka International Cancer Institute, Osaka, Osaka-shi
- Hospital Universitario Virgen del Rocio, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: No